CLINICAL TRIAL: NCT07041099
Title: A Phase 1b, Open-Label Study of CLN-978 for the Treatment of Active, Moderate to Severe Sjogren's Disease
Brief Title: A Study of CLN-978, a Subcutaneously Administered CD19-directed T Cell Engager, in Subjects With Sjogren's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cullinan Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN-978-SJ-101
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Sjögren; Sjogren Disease; Sjogren's Syndrome
Keywords: CLN-978
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A Dose Escalation (Experimental): Patients with Sjogren's Disease treated with CLN-978 in dose escalation cohorts
  Interventions: Drug: CLN-978
- Part B Further Dose Evaluation (Experimental): Further evaluation of CLN-978 treatment of patients with Sjogren's Disease
  Interventions: Drug: CLN-978

INTERVENTIONS:
Drug: CLN-978 — Specified dose on specified days

SUMMARY:
A phase 1b, open-label study of CLN-978 administered subcutaneously in patients with active, moderate to severe Sjogren's Disease.

ELIGIBILITY:
Inclusion

* Diagnosis of SjD at least 24 weeks prior to Screening Visit and meet the 2016 EULAR / ACR Classification Criteria for SjD at Screening.
* Have active moderate to severe disease (i.e., ESSDAI ≥5) at Screening.
* Laboratory parameters including the following:

  * Absolute lymphocyte count (ALC) ≥0.5 × 10^9/L
  * Peripheral CD19+ B cell count ≥25 cells/µL
  * Absolute neutrophil count (ANC) ≥1.0 × 10^9/L
  * Hemoglobin (Hgb) ≥8 g/dL
  * Platelet count ≥75 × 10^9/L
  * Total bilirubin ≤1.5 × ULN, except patients with confirmed Gilbert's Syndrome
  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.0 × ULN
  * Estimated glomerular filtration rate (eGFR) based on the CKD-EPI formula ≥30 mL/min/1.73 m2

Exclusion

* Concomitant rheumatological autoimmune disease
* Considered at high risk for thrombosis
* Rapidly progressive glomerulonephritis and/or urine protein/creatinine >3 mg/mg (339 mg/mmol).
* Active, severe central nervous system manifestations of SjD.
* History of stroke, seizure, dementia, Parkinson's disease, coordination movement disorder, cerebellar diseases, psychosis, paresis, aphasia, and any other neurologic disorder that the Investigator feels would put the patient at undue risk or confound study results.
* Evidence of hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), Epstein-Barr virus (EBV), or cytomegalovirus (CMV) infection.
* Primary immunodeficiency or history of recurrent infections.
* History of splenectomy.
* Live or attenuated vaccine within 28 days prior to the Screening Visit or during the Screening Period.
* Active, clinically significant bacterial, viral, fungal, mycobacterial, parasitic, or other infection, including severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, within 14 days prior to Day 1.
* Active or latent tuberculosis (TB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 48 weeks
  Incidence and severity of adverse events (AEs), serious AEs (SAEs), AEs of special interest (AESIs).

SECONDARY OUTCOMES:
To evaluate the PK of CLN-978 | 48 weeks
  Serum concentrations of CLN-978
Detection of anti-drug antibodies | 48 weeks
  Detection of anti-drug antibodies
Change from baseline in B lymphocyte cell numbers in peripheral blood | 48 weeks
  B lymphocyte cell numbers and change from baseline in peripheral blood

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Cullinan Investigative Site, Plano, Texas
  - Cullinan Investigative Site, Salt Lake City, Utah
- Cullinan Investigative Site, Erlangen, Germany